CLINICAL TRIAL: NCT00470587
Title: Advantageous Predictors of Acute Coronary Syndromes Evaluation (APACE) Study
Acronym: APACE
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: APACE
Record Dates: First submitted 2007-05-07; First posted 2007-05-08 (Estimated); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Myocardial Infarction; Angina, Unstable
Keywords: chest pain; myocardial infarction; unstable angina
MeSH Terms: conditions — Myocardial Infarction; Angina, Unstable; Chest Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — EDTA plasma, Heparin, Serum, Citrate
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The triage of patients with suspected acute coronary syndrome in the emergency room is a time-consuming diagnostic challenge. Therefore high sensitive early markers for myocardial damage are needed for more rapidly rule out of acute myocardial infarction (AMI) - especially for the first 3 to 4 hours after onset of chest pain in AMI ("troponin-blind" period).

Therefore we test the hypothesis that the use meticulous patient history and novel cardiac markers can provide a faster detection or exclusion of AMI in patients presenting with acute chest pain to the emergency department.

The prospective cohort study is designed to enrol patients presenting with acute chest pain at rest within the last 12 hours to the emergency department. Several blood samples for detection of the new markers will be drawn and compared with the gold standard for the diagnosis of AMI (high-sensitivity cardiac troponin T). All patients will be contacted by telephone at 3, 12, 24 and 60 months to determine functional status, major adverse cardiac events (death, myocardial infarction, coronary artery bypass grafting, percutaneous coronary intervention), and the results of cardiac examination (stress test, coronary angiography) if performed.

DETAILED DESCRIPTION:
Background: The triage of patients with suspected acute coronary syndrome in the emergency room is a time-consuming diagnostic challenge. Triage and management of patients with low probability of coronary artery disease often cause excessive hospital costs. Therefore high sensitive early markers for myocardial damage are needed for more rapidly rule out of acute myocardial infarction (AMI).

Cardiac troponins (T and I) are currently the gold standard for definitive AMI diagnosis due to their high sensitivity and specificity for detection of myocardial cell injury. Unfortunately, troponin is undetectable by current assays in peripheral blood within 3 to 4 hours after onset of chest pain in AMI ("troponin-blind" period).

New cardiac markers such as the novel high-sensitive troponin I/T, ischemia modified albumin and placental growth factor have demonstrated certain advantages compared to troponin such as high negative predictive value for AMI, earlier verifiability in peripheral blood and possible value as independent risk marker. However, clinical evaluation in a large cohort of unselected patients presenting to an emergency department is still lacking.

Aim: To test the hypothesis that the use meticulous patient history and novel cardiac markers (including high-sensitive troponin I/T, myeloperoxidase, ischemia modified albumin, placental growth factor) can provide a faster detection or exclusion of AMI in patients presenting with acute chest pain to the emergency department.

Patients and Methods: The prospective cohort study is designed to enrol unselected patients presenting with acute chest pain at rest within the last 12 hours to the emergency department. Several blood samples for detection of the new markers will be drawn (baseline, 1, 2, 3 and 6 hours) and compared with the gold standard for the diagnosis of AMI (high-sensitivity cardiac troponin T). Timing and treatment of patients are left to the discretion of the attending physician and will be performed according to the standard house routine of the hospital. All patients will be contacted by telephone at 6, 12, 24 and 60 months to determine functional status, major adverse cardiac events (death, myocardial infarction, coronary artery bypass grafting, percutaneous coronary intervention), and the results of cardiac examination (stress test, coronary angiography) if performed.

Expected results: It is our hypothesis that the use meticulous patient history and novel cardiac markers can improve the detection of AMI by providing an early diagnosis for AMI with a high negative predictive value within the "troponin-blind" period.

Significance: The earlier detection of myocardial necrosis in peripheral blood could help to rule out AMI more rapidly. In addition it will allow a more rapid diagnosis and appropriate therapy of AMI. This can lead to a significant improvement in patient management and a reduction of in-hospital costs.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the emergency department
* Typical angina pectoris or other thoracic sensations that are suspected to be caused by myocardial ischemia
* Symptoms at rest or minor exertion
* Onset of symptoms within the last 12 hours prior to presentation
* Written informed consent

Exclusion Criteria:

* Age < 18 years
* Cardiogenic shock
* Terminal kidney disease requiring regular dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the emergency department with typical angina pectoris or other thoracic sensations at rest or minor exertion that are suspected to be caused by myocardial ischemia. Onset of symptoms within the last 12 hours prior to presentation.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2006-04; Primary Completion 2025-03-02 (Actual); Study Completion 2025-12 (Actual)

PRIMARY OUTCOMES:
Diagnostic utility of various biomarkers, detailed patient's history and examination as well as ECG findings for the early diagnosis of acute myocardial infarction | at admission

CONTACTS AND LOCATIONS:
Overall Officials: Christian Mueller, MD, Principal Investigator — University Hospital of Basel
Locations (13):
- Masaryk University Brno, Brno, Czechia
- Emergency Department San Martino Hospital, Genova, Italy
- Medical University of Silesia, Zabrze, Poland
- Spain (3):
  - Hospital Clinic of Barcelona, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Clinico San Carlos, Madrid
- Switzerland (7):
  - University Hospital of Basel, Basel
  - Kantonsspital Baselland, Standort Bruderholz, Bottmingen
  - Kantonsspital Baselland, Standort Liestal, Liestal
  - Klinik St. Anna, Lucerne
  - Kantonsspital Olten, Olten
  - Spital Limmattal, Schlieren
  - Universitätsspital Zürich, Zurich

REFERENCES:
- [Derived] Lopez-Ayala P, Boeddinghaus J, Koechlin L, Bima P, Glaeser J, Spagnuolo CC, Crisanti L, Miro O, Martin-Sanchez FJ, Christ M, Wildi K, Piazza S, Nestelberger T, Gimenez MR, Gehrke J, Formambuh J, Kaplan E, Hure G, Breidthardt T, Giannitsis E, Lindahl B, Marber M, Mahfoud F, Strebel I, Mueller C; APACE and TRAPID-AMI investigators. Incremental Value of Cardiac Myosin-Binding Protein C for the Early Diagnosis of Acute Myocardial Infarction. J Am Coll Cardiol. 2025 Dec 23;86(25):2616-2632. doi: 10.1016/j.jacc.2025.09.008. Epub 2025 Nov 12. PMID 41222525
- [Derived] Dugar F, Lopez-Ayala P, Koechlin L, Bima P, Glaeser J, Spagnuolo C, Crisanti L, Wick C, Wildi K, Kaplan E, Strebel I, Miro O, Martin-Sanchez FJ, Christ M, Morawiec B, Gimenez MR, Nestelberger T, Boeddinghaus J, Mueller C; APACE investigators. Diagnostic and prognostic utility of endocan in suspected myocardial infarction: an international cohort study. Clin Chim Acta. 2026 Jan 1;578:120510. doi: 10.1016/j.cca.2025.120510. Epub 2025 Jul 25. PMID 40716696
- [Derived] Wildi K, Gimenez MR, Boeddinghaus J, Nestelberger T, Lopez-Ayala P, Koechlin L, Gerstenberger M, Carter N, Bima P, Glaeser J, Spagnuolo C, Miro O, Martin-Sanchez FJ, Christ M, Keller DI, Gualandro DM, Kawecki D, Rentsch K, Mahfoud F, Mueller C; APACE Investigators dagger. Possible Misdiagnosis of Myocardial Infarction Using Regulatory-Approved and Close-to-Bioequivalent Upper Limits of Normal for Cardiac Troponin. J Am Heart Assoc. 2025 May 20;14(10):e040468. doi: 10.1161/JAHA.124.040468. Epub 2025 May 13. PMID 40357766
- [Derived] Koechlin L, Boeddinghaus J, Lopez-Ayala P, Reber C, Nestelberger T, Wildi K, Spagnuolo CC, Strebel I, Glaeser J, Bima P, Crisanti L, Herraiz-Recuenco L, Dubach E, Miro O, Martin-Sanchez FJ, Kawecki D, Keller DI, Christ M, Buser A, Gimenez MR, Storvold GL, Broughton MN, Omland T, Lyngbakken MN, Rosjo H, Mueller C; APACE Investigators. Clinical and Analytical Performance of a Novel Point-of-Care High-Sensitivity Cardiac Troponin I Assay. J Am Coll Cardiol. 2024 Aug 20;84(8):726-740. doi: 10.1016/j.jacc.2024.05.056. PMID 39142727
- [Derived] Albus M, Zimmermann T, Median D, Rumora K, Isayeva G, Amrein M, Schaefer I, Walter J, Michel E, Hure G, Strebel I, Caobelli F, Haaf P, Frey SM, Mueller C, Zellweger MJ. Combining anatomical and biochemical markers in the detection and risk stratification of coronary artery disease. Eur Heart J Cardiovasc Imaging. 2024 Aug 26;25(9):1197-1205. doi: 10.1093/ehjci/jeae093. PMID 38591997
- [Derived] Boeddinghaus J, Doudesis D, Lopez-Ayala P, Lee KK, Koechlin L, Wildi K, Nestelberger T, Borer R, Miro O, Martin-Sanchez FJ, Strebel I, Rubini Gimenez M, Keller DI, Christ M, Bularga A, Li Z, Ferry AV, Tuck C, Anand A, Gray A, Mills NL, Mueller C; CoDE-ACS and APACE Investigators. Machine Learning for Myocardial Infarction Compared With Guideline-Recommended Diagnostic Pathways. Circulation. 2024 Apr 2;149(14):1090-1101. doi: 10.1161/CIRCULATIONAHA.123.066917. Epub 2024 Feb 12. PMID 38344871
- [Derived] Koechlin L, Boeddinghaus J, Lopez-Ayala P, Wildi K, Nestelberger T, Wussler D, Guzman Tacla CA, Holder T, Muench-Gerber T, Glaeser J, Sanchez AY, Miro O, Martin-Sanchez FJ, Kawecki D, Buergler F, Buser A, Hure G, Gimenez MR, Keller DI, Christ M, Mueller C; APACE investigators. External validation of the 0/1h-algorithm and derivation of a 0/2h-algorithm using a new point-of-care Hs-cTnI assay. Am Heart J. 2024 Feb;268:104-113. doi: 10.1016/j.ahj.2023.11.014. Epub 2023 Dec 1. PMID 38042459
- [Derived] Bima P, Lopez-Ayala P, Koechlin L, Boeddinghaus J, Nestelberger T, Okamura B, Muench-Gerber TS, Sanzone A, Skolozubova D, Djurdjevic D, Rubini Gimenez M, Wildi K, Miro O, Martinez-Nadal G, Martin-Sanchez FJ, Christ M, Keller D, Lindahl B, Giannitsis E, Mueller C; APACE and TRAPID-AMI Investigators. Chest Pain in Cancer Patients: Prevalence of Myocardial Infarction and Performance of High-Sensitivity Cardiac Troponins. JACC CardioOncol. 2023 Aug 26;5(5):591-609. doi: 10.1016/j.jaccao.2023.08.001. eCollection 2023 Oct. PMID 37969646
- [Derived] Yufera-Sanchez A, Lopez-Ayala P, Nestelberger T, Wildi K, Boeddinghaus J, Koechlin L, Rubini Gimenez M, Sakiz H, Bima P, Miro O, Martin-Sanchez FJ, Christ M, Keller DI, Gualandro DM, Kawecki D, Rentsch K, Buser A, Mueller C; APACE Investigators. Combining glucose and high-sensitivity cardiac troponin in the early diagnosis of acute myocardial infarction. Sci Rep. 2023 Sep 5;13(1):14598. doi: 10.1038/s41598-023-37093-1. PMID 37670005
- [Derived] Fernandez-Cisnal A, Lopez-Ayala P, Valero E, Koechlin L, Catarrala A, Boeddinghaus J, Noceda J, Nestelberger T, Miro O, Julio N, Mueller C, Sanchis J. Derivation and external validation of machine-learning models for risk stratification in chest pain with normal troponin. Eur Heart J Acute Cardiovasc Care. 2023 Nov 16;12(11):743-752. doi: 10.1093/ehjacc/zuad089. PMID 37531633
- [Derived] Meier M, Boeddinghaus J, Nestelberger T, Koechlin L, Lopez-Ayala P, Wussler D, Walter JE, Zimmermann T, Badertscher P, Wildi K, Gimenez MR, Puelacher C, Glarner N, Magni J, Miro O, Martin-Sanchez FJ, Kawecki D, Keller DI, Gualandro DM, Twerenbold R, Nickel CH, Bingisser R, Mueller C; APACE investigators. Comparing the utility of clinical risk scores and integrated clinical judgement in patients with suspected acute coronary syndrome. Eur Heart J Acute Cardiovasc Care. 2023 Oct 25;12(10):693-702. doi: 10.1093/ehjacc/zuad081. PMID 37435949
- [Derived] Boeddinghaus J, Nestelberger T, Koechlin L, Lopez-Ayala P, Wussler D, Mais M, Zwimpfer L, Zimmermann T, Wildi K, Gimenez MR, Strebel I, Miro O, Martin-Sanchez FJ, Parenica J, Keller DI, Gualandro DM, Nickel CH, Bingisser R, Christ M, Mueller C; APACE investigators. Association of accompanying dyspnoea with diagnosis and outcome of patients presenting with acute chest discomfort. Eur Heart J Acute Cardiovasc Care. 2023 May 4;12(5):283-295. doi: 10.1093/ehjacc/zuad026. PMID 36917461
- [Derived] Koechlin L, Strebel I, Zimmermann T, Nestelberger T, Walter J, Lopez-Ayala P, Boeddinghaus J, Shrestha S, Arslani K, Stefanelli S, Reuthebuch B, Wussler D, Ratmann PD, Christ M, Badertscher P, Wildi K, Gimenez MR, Gualandro DM, Miro O, Fuenzalida C, Martin-Sanchez FJ, Kawecki D, Burgler F, Keller DI, Abacherli R, Reuthebuch O, Eckstein FS, Twerenbold R, Reichlin T, Mueller C; APACE investigators. Hyperacute T Wave in the Early Diagnosis of Acute Myocardial Infarction. Ann Emerg Med. 2023 Aug;82(2):194-202. doi: 10.1016/j.annemergmed.2022.12.003. Epub 2023 Feb 10. PMID 36774205
- [Derived] Koechlin L, Boeddinghaus J, Lopez-Ayala P, Nestelberger T, Wussler D, Mais F, Twerenbold R, Zimmermann T, Wildi K, Koppen AM, Miro O, Martin-Sanchez FJ, Kawecki D, Geigy N, Keller DI, Christ M, Buser A, Gimenez MR, Bernasconi L, Hammerer-Lercher A, Mueller C; APACE investigators. Diagnostic discrimination of a novel high-sensitivity cardiac troponin I assay and derivation/validation of an assay-specific 0/1h-algorithm. Am Heart J. 2023 Jan;255:58-70. doi: 10.1016/j.ahj.2022.10.007. Epub 2022 Oct 13. PMID 36243111
- [Derived] Ratmann PD, Boeddinghaus J, Nestelberger T, Lopez-Ayala P, Hure G, Gehrke J, Koechlin L, Wildi K, Mueller P, Bima P, Wussler D, Gisler N, Miro O, Martin-Sanchez FJ, Christ M, Gualandro DM, Twerenbold R, Gimenez MR, Keller DI, Buser A, Mueller C; APACE Investigators. Extending the no objective testing rules to patients triaged by the European Society of Cardiology 0/1-hour algorithms. Eur Heart J Acute Cardiovasc Care. 2022 Nov 30;11(11):834-840. doi: 10.1093/ehjacc/zuac120. PMID 36179255
- [Derived] Koechlin L, Boeddinghaus J, Nestelberger T, Lopez-Ayala P, Shrestha S, Wussler D, Haeni N, Walter JE, Twerenbold R, Eckstein FS, Reuthebuch O, McCord J, Nowak RM, Christenson RH, deFilippi CR, Apple FS, Mueller C; APACE and High-US investigators. Lower diagnostic accuracy of hs-cTnI in patients with prior coronary artery bypass grafting. Int J Cardiol. 2022 May 1;354:1-6. doi: 10.1016/j.ijcard.2022.02.025. Epub 2022 Feb 18. PMID 35189168
- [Derived] Kaier TE, Twerenbold R, Lopez-Ayala P, Nestelberger T, Boeddinghaus J, Alaour B, Huber IM, Zhi Y, Koechlin L, Wussler D, Wildi K, Shrestha S, Strebel I, Miro O, Martin-Sanchez JF, Christ M, Kawecki D, Keller DI, Rubini Gimenez M, Marber M, Mueller C; APACE Investigators. A 0/1h-algorithm using cardiac myosin-binding protein C for early diagnosis of myocardial infarction. Eur Heart J Acute Cardiovasc Care. 2022 Jun 7;11(4):325-335. doi: 10.1093/ehjacc/zuac007. PMID 35149868
- [Derived] Prepoudis A, Koechlin L, Nestelberger T, Boeddinghaus J, Lopez-Ayala P, Wussler D, Zimmermann T, Rubini Gimenez M, Strebel I, Puelacher C, Shrestha S, Keller DI, Christ M, Gualandro DM, Twerenbold R, Martinez-Nadal G, Lopez-Barbeito B, Miro O, Mueller C; APACE investigators. Incidence, clinical presentation, management, and outcome of acute pericarditis and myopericarditis. Eur Heart J Acute Cardiovasc Care. 2022 Feb 8;11(2):137-147. doi: 10.1093/ehjacc/zuab108. PMID 34849666
- [Derived] Koechlin L, Boeddinghaus J, Nestelberger T, Lopez-Ayala P, Wussler D, Shrestha S, Resa T, Wildi K, Bakula A, Frey S, Miro O, Martin-Sanchez FJ, Strebel I, Gualandro DM, Eckstein FS, Reuthebuch O, Keller DI, Twerenbold R, Gimenez MR, Mueller C; APACE investigators. Performance of the ESC 0/2h-algorithm using high-sensitivity cardiac troponin I in the early diagnosis of myocardial infarction. Am Heart J. 2021 Dec;242:132-137. doi: 10.1016/j.ahj.2021.08.008. Epub 2021 Sep 9. PMID 34508692
- [Derived] Boeddinghaus J, Lopez-Ayala P, Nestelberger T, Koechlin L, Munch T, Miro O, Gimenez MR, Mueller C; APACE Investigators. Prospective Validation of the ESC 0/1h-Algorithm Using High-Sensitivity Cardiac Troponin I. Am J Cardiol. 2021 Nov 1;158:152-153. doi: 10.1016/j.amjcard.2021.08.007. Epub 2021 Aug 30. No abstract available. PMID 34470703
- [Derived] Lopez-Ayala P, Nestelberger T, Boeddinghaus J, Koechlin L, Ratmann PD, Strebel I, Gehrke J, Meier S, Walter J, Rubini Gimenez M, Mutschler E, Miro O, Lopez-Barbeito B, Martin-Sanchez FJ, Rodriguez-Adrada E, Keller DI, Newby LK, Twerenbold R, Giannitsis E, Lindahl B, Mueller C; APACE and TRAPID-AMI Investigatorsdagger. Novel Criteria for the Observe-Zone of the ESC 0/1h-hs-cTnT Algorithm. Circulation. 2021 Sep 7;144(10):773-787. doi: 10.1161/CIRCULATIONAHA.120.052982. Epub 2021 Aug 11. PMID 34376064
- [Derived] Nestelberger T, Boeddinghaus J, Gimenez MR, Lopez-Ayala P, Ratmann PD, Badertscher P, Wildi K, Wussler D, Koechlin L, Arslani K, Zimmermann T, Freese M, Rinderknecht T, Miro O, Martin-Sanchez FJ, Kawecki D, Geigy N, Keller D, Twerenbold R, Muller C; APACE investigators. Direct comparison of high-sensitivity cardiac troponin T and I in the early differentiation of type 1 vs. type 2 myocardial infarction. Eur Heart J Acute Cardiovasc Care. 2022 Jan 12;11(1):62-74. doi: 10.1093/ehjacc/zuab039. PMID 34195803
- [Derived] Boeddinghaus J, Nestelberger T, Lopez-Ayala P, Koechlin L, Buechi M, Miro O, Keller DI, Gimenez MR, Twerenbold R, Mueller C; APACE Investigators. Diagnostic Performance of the European Society of Cardiology 0/1-h Algorithms in Late Presenters. J Am Coll Cardiol. 2021 Mar 9;77(9):1264-1267. doi: 10.1016/j.jacc.2021.01.004. No abstract available. PMID 33663745
- [Derived] Koechlin L, Boeddinghaus J, Nestelberger T, Miro O, Fuenzalida C, Martinez-Nadal G, Lopez B, Wussler D, Walter J, Zimmermann T, Troester V, Lopez-Ayala P, Baumgartner B, Ratmann PD, Diebold M, Prepoudis A, Huber J, Christ M, Wildi K, Rubini Gimenez M, Strebel I, Gualandro DM, Martin-Sanchez FJ, Kawecki D, Keller DI, Reuthebuch O, Eckstein FS, Reichlin T, Twerenbold R, Mueller C; APACE investigators. Clinical presentation of patients with prior coronary artery bypass grafting and suspected acute myocardial infarction. Eur Heart J Acute Cardiovasc Care. 2021 Oct 1;10(7):746-755. doi: 10.1093/ehjacc/zuaa020. PMID 33620434
- [Derived] Troester V, Strebel I, Nestelberger T, Boeddinghaus J, Rubini Gimenez M, Lopez-Ayala P, Koechlin L, Glarner N, Prepoudis A, Miro O, Martin-Sanchez FJ, Kawecki D, Keller DI, Twerenbold R, Mueller C; APACE Investigators *. Association of Previous Myocardial Infarction and Time to Presentation With Suspected Acute Myocardial Infarction. J Am Heart Assoc. 2021 Jan 5;10(1):e017829. doi: 10.1161/JAHA.120.017829. Epub 2020 Dec 26. No abstract available. PMID 33356355
- [Derived] Rubini Gimenez M, Wildi K, Wussler D, Koechlin L, Boeddinghaus J, Nestelberger T, Badertscher P, Sedlmayer R, Puelacher C, Zimmermann T, du Fay de Lavallaz J, Lopez-Ayala P, Leu K, Rentsch K, Miro O, Lopez B, Martin-Sanchez FJ, Bustamante J, Kawecki D, Parenica J, Lohrmann J, Kloos W, Buser A, Keller DI, Reichlin T, Twerenbold R, Mueller C. Early kinetics of cardiac troponin in suspected acute myocardial infarction. Rev Esp Cardiol (Engl Ed). 2021 Jun;74(6):502-509. doi: 10.1016/j.rec.2020.04.008. Epub 2020 May 22. English, Spanish. PMID 32451223
- [Derived] Boeddinghaus J, Nestelberger T, Koechlin L, Wussler D, Lopez-Ayala P, Walter JE, Troester V, Ratmann PD, Seidel F, Zimmermann T, Badertscher P, Wildi K, Rubini Gimenez M, Potlukova E, Strebel I, Freese M, Miro O, Martin-Sanchez FJ, Kawecki D, Keller DI, Gualandro DM, Christ M, Twerenbold R, Mueller C; APACE Investigators. Early Diagnosis of Myocardial Infarction With Point-of-Care High-Sensitivity Cardiac Troponin I. J Am Coll Cardiol. 2020 Mar 17;75(10):1111-1124. doi: 10.1016/j.jacc.2019.12.065. PMID 32164884
- [Derived] Haller PM, Boeddinghaus J, Neumann JT, Sorensen NA, Hartikainen TS, Gossling A, Nestelberger T, Twerenbold R, Lehmacher J, Keller T, Zeller T, Blankenberg S, Mueller C, Westermann D. Performance of the ESC 0/1-h and 0/3-h Algorithm for the Rapid Identification of Myocardial Infarction Without ST-Elevation in Patients With Diabetes. Diabetes Care. 2020 Feb;43(2):460-467. doi: 10.2337/dc19-1327. Epub 2019 Dec 16. PMID 31843947
- [Derived] Nestelberger T, Boeddinghaus J, Greenslade J, Parsonage WA, Than M, Wussler D, Lopez-Ayala P, Zimmermann T, Meier M, Troester V, Badertscher P, Koechlin L, Wildi K, Anwar M, Freese M, Keller DI, Reichlin T, Twerenbold R, Cullen L, Mueller C; APACE and ADAPT Investigators. Two-Hour Algorithm for Rapid Triage of Suspected Acute Myocardial Infarction Using a High-Sensitivity Cardiac Troponin I Assay. Clin Chem. 2019 Nov;65(11):1437-1447. doi: 10.1373/clinchem.2019.305193. Epub 2019 Sep 30. PMID 31570634
- [Derived] Boeddinghaus J, Twerenbold R, Nestelberger T, Koechlin L, Wussler D, Meier M, Troester V, Zimmermann T, Badertscher P, Wildi K, Rubini Gimenez M, Lopez-Ayala P, Potlukova E, Miro O, Martin-Sanchez FJ, Kawecki D, Geigy N, Keller DI, Reichlin T, Mueller C; APACE investigators. Clinical Use of a New High-Sensitivity Cardiac Troponin I Assay in Patients with Suspected Myocardial Infarction. Clin Chem. 2019 Nov;65(11):1426-1436. doi: 10.1373/clinchem.2019.304725. Epub 2019 Sep 30. PMID 31570633
- [Derived] Nestelberger T, Boeddinghaus J, Wussler D, Twerenbold R, Badertscher P, Wildi K, Miro O, Lopez B, Martin-Sanchez FJ, Muzyk P, Koechlin L, Baumgartner B, Meier M, Troester V, Rubini Gimenez M, Puelacher C, du Fay de Lavallaz J, Walter J, Kozhuharov N, Zimmermann T, Gualandro DM, Michou E, Potlukova E, Geigy N, Keller DI, Reichlin T, Mueller C; APACE Investigators. Predicting Major Adverse Events in Patients With Acute Myocardial Infarction. J Am Coll Cardiol. 2019 Aug 20;74(7):842-854. doi: 10.1016/j.jacc.2019.06.025. PMID 31416527
- [Derived] Neumann JT, Twerenbold R, Ojeda F, Sorensen NA, Chapman AR, Shah ASV, Anand A, Boeddinghaus J, Nestelberger T, Badertscher P, Mokhtari A, Pickering JW, Troughton RW, Greenslade J, Parsonage W, Mueller-Hennessen M, Gori T, Jernberg T, Morris N, Liebetrau C, Hamm C, Katus HA, Munzel T, Landmesser U, Salomaa V, Iacoviello L, Ferrario MM, Giampaoli S, Kee F, Thorand B, Peters A, Borchini R, Jorgensen T, Soderberg S, Sans S, Tunstall-Pedoe H, Kuulasmaa K, Renne T, Lackner KJ, Worster A, Body R, Ekelund U, Kavsak PA, Keller T, Lindahl B, Wild P, Giannitsis E, Than M, Cullen LA, Mills NL, Mueller C, Zeller T, Westermann D, Blankenberg S; COMPASS-MI Study Group. Application of High-Sensitivity Troponin in Suspected Myocardial Infarction. N Engl J Med. 2019 Jun 27;380(26):2529-2540. doi: 10.1056/NEJMoa1803377. PMID 31242362
- [Derived] Nestelberger T, Cullen L, Lindahl B, Reichlin T, Greenslade JH, Giannitsis E, Christ M, Morawiec B, Miro O, Martin-Sanchez FJ, Wussler DN, Koechlin L, Twerenbold R, Parsonage W, Boeddinghaus J, Rubini Gimenez M, Puelacher C, Wildi K, Buerge T, Badertscher P, DuFaydeLavallaz J, Strebel I, Croton L, Bendig G, Osswald S, Pickering JW, Than M, Mueller C; APACE, ADAPT and TRAPID-AMI Investigators. Diagnosis of acute myocardial infarction in the presence of left bundle branch block. Heart. 2019 Oct;105(20):1559-1567. doi: 10.1136/heartjnl-2018-314673. Epub 2019 May 29. PMID 31142594
- [Derived] Hillinger P, Strebel I, Abacherli R, Twerenbold R, Wildi K, Bernhard D, Nestelberger T, Boeddinghaus J, Badertscher P, Wussler D, Koechlin L, Zimmermann T, Puelacher C, Rubini Gimenez M, du Fay de Lavallaz J, Walter J, Geigy N, Keller DI, Reichlin T, Mueller C; APACE Investigators. Prospective validation of current quantitative electrocardiographic criteria for ST-elevation myocardial infarction. Int J Cardiol. 2019 Oct 1;292:1-12. doi: 10.1016/j.ijcard.2019.04.041. Epub 2019 Apr 11. PMID 31056411
- [Derived] Boeddinghaus J, Nestelberger T, Twerenbold R, Koechlin L, Meier M, Troester V, Wussler D, Badertscher P, Wildi K, Puelacher C, du Fay de Lavallaz J, Rubini Gimenez M, Zimmermann T, Hafner B, Potlukova E, Miro O, Martin-Sanchez FJ, Keller DI, Reichlin T, Mueller C; APACE investigators. High-Sensitivity Cardiac Troponin I Assay for Early Diagnosis of Acute Myocardial Infarction. Clin Chem. 2019 Jul;65(7):893-904. doi: 10.1373/clinchem.2018.300061. Epub 2019 Apr 15. PMID 30988172
- [Derived] Morawiec B, Boeddinghaus J, Wussler D, Badertscher P, Koechlin L, Metry F, Twerenbold R, Nestelberger T, Kawecki D, Mueller C; APACE Investigators. Modified HEART Score and High-Sensitivity Cardiac Troponin in Patients With Suspected Acute Myocardial Infarction. J Am Coll Cardiol. 2019 Feb 26;73(7):873-875. doi: 10.1016/j.jacc.2018.12.013. No abstract available. PMID 30784680
- [Derived] Wildi K, Nestelberger T, Wussler D, Boeddinghaus J, Badertscher P, Koechlin L, Duwe P, Rubini Gimenez M, Twerenbold R, Mueller C. Impact of Food and Drug Administration Regulatory Approach on the 0/2-Hour Algorithm for Rapid Triage of Suspected Myocardial Infarction. Circ Cardiovasc Qual Outcomes. 2019 Jan;12(1):e005188. doi: 10.1161/CIRCOUTCOMES.118.005188. No abstract available. PMID 30630358
- [Derived] Boeddinghaus J, Nestelberger T, Badertscher P, Twerenbold R, Fitze B, Wussler D, Strebel I, Rubini Gimenez M, Wildi K, Puelacher C, du Fay de Lavallaz J, Oehen L, Walter J, Miro O, Martin-Sanchez FJ, Morawiec B, Potlukova E, Keller DI, Reichlin T, Mueller C; APACE Investigators. Predicting Acute Myocardial Infarction with a Single Blood Draw. Clin Chem. 2019 Mar;65(3):437-450. doi: 10.1373/clinchem.2018.294124. Epub 2019 Jan 9. PMID 30626633
- [Derived] Wildi K, Boeddinghaus J, Nestelberger T, Twerenbold R, Badertscher P, Wussler D, Gimenez MR, Puelacher C, du Fay de Lavallaz J, Dietsche S, Walter J, Kozhuharov N, Morawiec B, Miro O, Javier Martin-Sanchez F, Subramaniam S, Geigy N, Keller DI, Reichlin T, Mueller C; APACE investigators. Comparison of fourteen rule-out strategies for acute myocardial infarction. Int J Cardiol. 2019 May 15;283:41-47. doi: 10.1016/j.ijcard.2018.11.140. Epub 2018 Dec 3. PMID 30545622
- [Derived] Boeddinghaus J, Nestelberger T, Twerenbold R, Neumann JT, Lindahl B, Giannitsis E, Sorensen NA, Badertscher P, Jann JE, Wussler D, Puelacher C, Rubini Gimenez M, Wildi K, Strebel I, Du Fay de Lavallaz J, Selman F, Sabti Z, Kozhuharov N, Potlukova E, Rentsch K, Miro O, Martin-Sanchez FJ, Morawiec B, Parenica J, Lohrmann J, Kloos W, Buser A, Geigy N, Keller DI, Osswald S, Reichlin T, Westermann D, Blankenberg S, Mueller C; APACE, BACC, and TRAPID-AMI Investigators. Impact of age on the performance of the ESC 0/1h-algorithms for early diagnosis of myocardial infarction. Eur Heart J. 2018 Nov 7;39(42):3780-3794. doi: 10.1093/eurheartj/ehy514. PMID 30169752
- [Derived] Boeddinghaus J, Twerenbold R, Nestelberger T, Badertscher P, Wildi K, Puelacher C, du Fay de Lavallaz J, Keser E, Rubini Gimenez M, Wussler D, Kozhuharov N, Rentsch K, Miro O, Martin-Sanchez FJ, Morawiec B, Stefanelli S, Geigy N, Keller DI, Reichlin T, Mueller C; APACE Investigators. Clinical Validation of a Novel High-Sensitivity Cardiac Troponin I Assay for Early Diagnosis of Acute Myocardial Infarction. Clin Chem. 2018 Sep;64(9):1347-1360. doi: 10.1373/clinchem.2018.286906. Epub 2018 Jun 25. PMID 29941469
- [Derived] Wildi K, Singeisen H, Twerenbold R, Badertscher P, Wussler D, Klinkenberg LJJ, Meex SJR, Nestelberger T, Boeddinghaus J, Miro O, Martin-Sanchez FJ, Morawiec B, Muzyk P, Parenica J, Keller DI, Geigy N, Potlukova E, Sabti Z, Kozhuharov N, Puelacher C, du Fay de Lavallaz J, Rubini Gimenez M, Shrestha S, Marzano G, Rentsch K, Osswald S, Reichlin T, Mueller C; APACE Investigators. Circadian rhythm of cardiac troponin I and its clinical impact on the diagnostic accuracy for acute myocardial infarction. Int J Cardiol. 2018 Nov 1;270:14-20. doi: 10.1016/j.ijcard.2018.05.136. Epub 2018 Jun 4. PMID 29891238
- [Derived] van der Linden N, Wildi K, Twerenbold R, Pickering JW, Than M, Cullen L, Greenslade J, Parsonage W, Nestelberger T, Boeddinghaus J, Badertscher P, Rubini Gimenez M, Klinkenberg LJJ, Bekers O, Schoni A, Keller DI, Sabti Z, Puelacher C, Cupa J, Schumacher L, Kozhuharov N, Grimm K, Shrestha S, Flores D, Freese M, Stelzig C, Strebel I, Miro O, Rentsch K, Morawiec B, Kawecki D, Kloos W, Lohrmann J, Richards AM, Troughton R, Pemberton C, Osswald S, van Dieijen-Visser MP, Mingels AM, Reichlin T, Meex SJR, Mueller C. Combining High-Sensitivity Cardiac Troponin I and Cardiac Troponin T in the Early Diagnosis of Acute Myocardial Infarction. Circulation. 2018 Sep 4;138(10):989-999. doi: 10.1161/CIRCULATIONAHA.117.032003. PMID 29691270
- [Derived] Rubini Gimenez M, Badertscher P, Twerenbold R, Boeddinghaus J, Nestelberger T, Wussler D, Miro O, Martin-Sanchez FJ, Reichlin T, Mueller C. Impact of the US Food and Drug Administration-Approved Sex-Specific Cutoff Values for High-Sensitivity Cardiac Troponin T to Diagnose Myocardial Infarction. Circulation. 2018 Apr 24;137(17):1867-1869. doi: 10.1161/CIRCULATIONAHA.117.031940. No abstract available. PMID 29685935
- [Derived] Badertscher P, Boeddinghaus J, Nestelberger T, Twerenbold R, Wildi K, Sabti Z, Puelacher C, Rubini Gimenez M, Pfaffli J, Flores D, du Fay de Lavallaz J, Miro O, Martin-Sanchez FJ, Morawiec B, Lohrmann J, Buser A, Keller DI, Geigy N, Reichlin T, Mueller C. Effect of Acute Coronary Syndrome Probability on Diagnostic and Prognostic Performance of High-Sensitivity Cardiac Troponin. Clin Chem. 2018 Mar;64(3):515-525. doi: 10.1373/clinchem.2017.279513. Epub 2018 Jan 17. PMID 29343534
- [Derived] Twerenbold R, Badertscher P, Boeddinghaus J, Nestelberger T, Wildi K, Puelacher C, Sabti Z, Rubini Gimenez M, Tschirky S, du Fay de Lavallaz J, Kozhuharov N, Sazgary L, Mueller D, Breidthardt T, Strebel I, Flores Widmer D, Shrestha S, Miro O, Martin-Sanchez FJ, Morawiec B, Parenica J, Geigy N, Keller DI, Rentsch K, von Eckardstein A, Osswald S, Reichlin T, Mueller C. 0/1-Hour Triage Algorithm for Myocardial Infarction in Patients With Renal Dysfunction. Circulation. 2018 Jan 30;137(5):436-451. doi: 10.1161/CIRCULATIONAHA.117.028901. Epub 2017 Nov 3. PMID 29101287
- [Derived] Kaier TE, Twerenbold R, Puelacher C, Marjot J, Imambaccus N, Boeddinghaus J, Nestelberger T, Badertscher P, Sabti Z, Gimenez MR, Wildi K, Hillinger P, Grimm K, Loeffel S, Shrestha S, Widmer DF, Cupa J, Kozhuharov N, Miro O, Martin-Sanchez FJ, Morawiec B, Rentsch K, Lohrmann J, Kloos W, Osswald S, Reichlin T, Weber E, Marber M, Mueller C. Direct Comparison of Cardiac Myosin-Binding Protein C With Cardiac Troponins for the Early Diagnosis of Acute Myocardial Infarction. Circulation. 2017 Oct 17;136(16):1495-1508. doi: 10.1161/CIRCULATIONAHA.117.028084. Epub 2017 Sep 26. PMID 28972002
- [Derived] Nestelberger T, Boeddinghaus J, Badertscher P, Twerenbold R, Wildi K, Breitenbucher D, Sabti Z, Puelacher C, Rubini Gimenez M, Kozhuharov N, Strebel I, Sazgary L, Schneider D, Jann J, du Fay de Lavallaz J, Miro O, Martin-Sanchez FJ, Morawiec B, Kawecki D, Muzyk P, Keller DI, Geigy N, Osswald S, Reichlin T, Mueller C; APACE Investigators. Effect of Definition on Incidence and Prognosis of Type 2 Myocardial Infarction. J Am Coll Cardiol. 2017 Sep 26;70(13):1558-1568. doi: 10.1016/j.jacc.2017.07.774. PMID 28935032
- [Derived] Twerenbold R, Badertscher P, Boeddinghaus J, Nestelberger T, Wildi K, Rubini Gimenez M, Miro O, Martin-Sanchez FJ, Reichlin T, Mueller C. Effect of the FDA Regulatory Approach on the 0/1-h Algorithm for Rapid Diagnosis of MI. J Am Coll Cardiol. 2017 Sep 19;70(12):1532-1534. doi: 10.1016/j.jacc.2017.07.746. No abstract available. PMID 28911517
- [Derived] Wildi K, Cullen L, Twerenbold R, Greenslade JH, Parsonage W, Boeddinghaus J, Nestelberger T, Sabti Z, Rubini-Gimenez M, Puelacher C, Cupa J, Schumacher L, Badertscher P, Grimm K, Kozhuharov N, Stelzig C, Freese M, Rentsch K, Lohrmann J, Kloos W, Buser A, Reichlin T, Pickering JW, Than M, Mueller C. Direct Comparison of 2 Rule-Out Strategies for Acute Myocardial Infarction: 2-h Accelerated Diagnostic Protocol vs 2-h Algorithm. Clin Chem. 2017 Jul;63(7):1227-1236. doi: 10.1373/clinchem.2016.268359. Epub 2017 May 17. PMID 28515106
- [Derived] Boeddinghaus J, Nestelberger T, Twerenbold R, Wildi K, Badertscher P, Cupa J, Burge T, Machler P, Corbiere S, Grimm K, Gimenez MR, Puelacher C, Shrestha S, Flores Widmer D, Fuhrmann J, Hillinger P, Sabti Z, Honegger U, Schaerli N, Kozhuharov N, Rentsch K, Miro O, Lopez B, Martin-Sanchez FJ, Rodriguez-Adrada E, Morawiec B, Kawecki D, Ganovska E, Parenica J, Lohrmann J, Kloos W, Buser A, Geigy N, Keller DI, Osswald S, Reichlin T, Mueller C. Direct Comparison of 4 Very Early Rule-Out Strategies for Acute Myocardial Infarction Using High-Sensitivity Cardiac Troponin I. Circulation. 2017 Apr 25;135(17):1597-1611. doi: 10.1161/CIRCULATIONAHA.116.025661. Epub 2017 Mar 10. PMID 28283497
- [Derived] Klinkenberg LJ, Wildi K, van der Linden N, Kouw IW, Niens M, Twerenbold R, Rubini Gimenez M, Puelacher C, Daniel Neuhaus J, Hillinger P, Nestelberger T, Boeddinghaus J, Grimm K, Sabti Z, Bons JA, van Suijlen JD, Tan FE, Ten Kate J, Bekers O, van Loon LJ, van Dieijen-Visser MP, Mueller C, Meex SJ. Diurnal Rhythm of Cardiac Troponin: Consequences for the Diagnosis of Acute Myocardial Infarction. Clin Chem. 2016 Dec;62(12):1602-1611. doi: 10.1373/clinchem.2016.257485. Epub 2016 Oct 5. PMID 27707754
- [Derived] Hillinger P, Twerenbold R, Wildi K, Rubini Gimenez M, Jaeger C, Boeddinghaus J, Nestelberger T, Grimm K, Reichlin T, Stallone F, Puelacher C, Sabti Z, Kozhuharov N, Honegger U, Ballarino P, Miro O, Denhaerynck K, Ekrem T, Kohler C, Bingisser R, Osswald S, Mueller C. Gender-specific uncertainties in the diagnosis of acute coronary syndrome. Clin Res Cardiol. 2017 Jan;106(1):28-37. doi: 10.1007/s00392-016-1020-y. Epub 2016 Jul 12. PMID 27406787
- [Derived] Twerenbold R, Jaeger C, Rubini Gimenez M, Wildi K, Reichlin T, Nestelberger T, Boeddinghaus J, Grimm K, Puelacher C, Moehring B, Pretre G, Schaerli N, Campodarve I, Rentsch K, Steuer S, Osswald S, Mueller C. Impact of high-sensitivity cardiac troponin on use of coronary angiography, cardiac stress testing, and time to discharge in suspected acute myocardial infarction. Eur Heart J. 2016 Nov 21;37(44):3324-3332. doi: 10.1093/eurheartj/ehw232. Epub 2016 Jun 29. PMID 27357358
- [Derived] Parsonage WA, Mueller C, Greenslade JH, Wildi K, Pickering J, Than M, Aldous S, Boeddinghaus J, Hammett CJ, Hawkins T, Nestelberger T, Reichlin T, Reidt S, Rubin Gimenez M, Tate JR, Twerenbold R, Ungerer JP, Cullen L. Validation of NICE diagnostic guidance for rule out of myocardial infarction using high-sensitivity troponin tests. Heart. 2016 Aug 15;102(16):1279-86. doi: 10.1136/heartjnl-2016-309270. Epub 2016 Jun 10. PMID 27288278
- [Derived] Abacherli R, Isaksen J, Schmid R, Leber R, Schmid HJ, Generali G. Digital DC-Reconstruction of AC-Coupled Electrophysiological Signals with a Single Inverting Filter. PLoS One. 2016 Mar 3;11(3):e0150207. doi: 10.1371/journal.pone.0150207. eCollection 2016. PMID 26938769
- [Derived] Hillinger P, Twerenbold R, Jaeger C, Wildi K, Reichlin T, Rubini Gimenez M, Engels U, Miro O, Boeddinghaus J, Puelacher C, Nestelberger T, Rothlisberger M, Ernst S, Rentsch K, Mueller C. Optimizing Early Rule-Out Strategies for Acute Myocardial Infarction: Utility of 1-Hour Copeptin. Clin Chem. 2015 Dec;61(12):1466-74. doi: 10.1373/clinchem.2015.242743. Epub 2015 Aug 31. PMID 26323282
- [Derived] Twerenbold R, Wildi K, Jaeger C, Gimenez MR, Reiter M, Reichlin T, Walukiewicz A, Gugala M, Krivoshei L, Marti N, Moreno Weidmann Z, Hillinger P, Puelacher C, Rentsch K, Honegger U, Schumacher C, Zurbriggen F, Freese M, Stelzig C, Campodarve I, Bassetti S, Osswald S, Mueller C. Optimal Cutoff Levels of More Sensitive Cardiac Troponin Assays for the Early Diagnosis of Myocardial Infarction in Patients With Renal Dysfunction. Circulation. 2015 Jun 9;131(23):2041-50. doi: 10.1161/CIRCULATIONAHA.114.014245. Epub 2015 May 6. PMID 25948542
- [Derived] Wildi K, Gimenez MR, Twerenbold R, Reichlin T, Jaeger C, Heinzelmann A, Arnold C, Nelles B, Druey S, Haaf P, Hillinger P, Schaerli N, Kreutzinger P, Tanglay Y, Herrmann T, Moreno Weidmann Z, Krivoshei L, Freese M, Stelzig C, Puelacher C, Rentsch K, Osswald S, Mueller C. Misdiagnosis of Myocardial Infarction Related to Limitations of the Current Regulatory Approach to Define Clinical Decision Values for Cardiac Troponin. Circulation. 2015 Jun 9;131(23):2032-40. doi: 10.1161/CIRCULATIONAHA.114.014129. Epub 2015 May 6. PMID 25948541
- [Derived] Reichlin T, Twerenbold R, Wildi K, Gimenez MR, Bergsma N, Haaf P, Druey S, Puelacher C, Moehring B, Freese M, Stelzig C, Krivoshei L, Hillinger P, Jager C, Herrmann T, Kreutzinger P, Radosavac M, Weidmann ZM, Pershyna K, Honegger U, Wagener M, Vuillomenet T, Campodarve I, Bingisser R, Miro O, Rentsch K, Bassetti S, Osswald S, Mueller C. Prospective validation of a 1-hour algorithm to rule-out and rule-in acute myocardial infarction using a high-sensitivity cardiac troponin T assay. CMAJ. 2015 May 19;187(8):E243-E252. doi: 10.1503/cmaj.141349. Epub 2015 Apr 13. PMID 25869867
- [Derived] Rubini Gimenez M, Twerenbold R, Jaeger C, Schindler C, Puelacher C, Wildi K, Reichlin T, Haaf P, Merk S, Honegger U, Wagener M, Druey S, Schumacher C, Krivoshei L, Hillinger P, Herrmann T, Campodarve I, Rentsch K, Bassetti S, Osswald S, Mueller C. One-hour rule-in and rule-out of acute myocardial infarction using high-sensitivity cardiac troponin I. Am J Med. 2015 Aug;128(8):861-870.e4. doi: 10.1016/j.amjmed.2015.01.046. Epub 2015 Mar 31. PMID 25840034
- [Derived] Wildi K, Cuculi F, Twerenbold R, Marxer T, Rubini Gimenez M, Reichlin T, Haaf P, Monsch R, Marsch S, Hunziker P, Bingisser R, Osswald S, Erne P, Mueller C. Incidence and timing of serious arrhythmias after early revascularization in non ST-elevation myocardial infarction. Eur Heart J Acute Cardiovasc Care. 2015 Aug;4(4):359-64. doi: 10.1177/2048872614557230. Epub 2014 Oct 27. PMID 25348273
- [Derived] Rubini Gimenez M, Reiter M, Twerenbold R, Reichlin T, Wildi K, Haaf P, Wicki K, Zellweger C, Hoeller R, Moehring B, Sou SM, Mueller M, Denhaerynck K, Meller B, Stallone F, Henseler S, Bassetti S, Geigy N, Osswald S, Mueller C. Sex-specific chest pain characteristics in the early diagnosis of acute myocardial infarction. JAMA Intern Med. 2014 Feb 1;174(2):241-9. doi: 10.1001/jamainternmed.2013.12199. PMID 24275751
- [Derived] Rubini Gimenez M, Hoeller R, Reichlin T, Zellweger C, Twerenbold R, Reiter M, Moehring B, Wildi K, Mosimann T, Mueller M, Meller B, Hochgruber T, Ziller R, Sou SM, Murray K, Sakarikos K, Ernst S, Gea J, Campodarve I, Vilaplana C, Haaf P, Steuer S, Minners J, Osswald S, Mueller C. Rapid rule out of acute myocardial infarction using undetectable levels of high-sensitivity cardiac troponin. Int J Cardiol. 2013 Oct 9;168(4):3896-901. doi: 10.1016/j.ijcard.2013.06.049. Epub 2013 Jul 20. PMID 23876467
- [Derived] Balmelli C, Meune C, Twerenbold R, Reichlin T, Rieder S, Drexler B, Rubini MG, Mosimann T, Reiter M, Haaf P, Mueller M, Ernst S, Ballarino P, Alafify AA, Zellweger C, Wildi K, Moehring B, Vilaplana C, Bernhard D, Merk S, Ebmeyer S, Freidank H, Osswald S, Mueller C. Comparison of the performances of cardiac troponins, including sensitive assays, and copeptin in the diagnostic of acute myocardial infarction and long-term prognosis between women and men. Am Heart J. 2013 Jul;166(1):30-7. doi: 10.1016/j.ahj.2013.03.014. Epub 2013 Apr 30. PMID 23816018
- [Derived] Hoeller R, Rubini Gimenez M, Reichlin T, Twerenbold R, Zellweger C, Moehring B, Wildi K, Freese M, Stelzig C, Hartmann B, Stoll M, Mosimann T, Reiter M, Haaf P, Mueller M, Meller B, Hochgruber T, Balmelli C, Sou SM, Murray K, Freidank H, Steuer S, Minners J, Osswald S, Mueller C. Normal presenting levels of high-sensitivity troponin and myocardial infarction. Heart. 2013 Nov;99(21):1567-72. doi: 10.1136/heartjnl-2013-303643. Epub 2013 Apr 19. PMID 23604180
- [Derived] Cullen L, Mueller C, Parsonage WA, Wildi K, Greenslade JH, Twerenbold R, Aldous S, Meller B, Tate JR, Reichlin T, Hammett CJ, Zellweger C, Ungerer JPJ, Rubini Gimenez M, Troughton R, Murray K, Brown AFT, Mueller M, George P, Mosimann T, Flaws DF, Reiter M, Lamanna A, Haaf P, Pemberton CJ, Richards AM, Chu K, Reid CM, Peacock WF, Jaffe AS, Florkowski C, Deely JM, Than M. Validation of high-sensitivity troponin I in a 2-hour diagnostic strategy to assess 30-day outcomes in emergency department patients with possible acute coronary syndrome. J Am Coll Cardiol. 2013 Oct 1;62(14):1242-1249. doi: 10.1016/j.jacc.2013.02.078. Epub 2013 Apr 10. PMID 23583250
- [Derived] Reichlin T, Twerenbold R, Maushart C, Reiter M, Moehring B, Schaub N, Balmelli C, Rubini Gimenez M, Hoeller R, Sakarikos K, Drexler B, Haaf P, Osswald S, Mueller C. Risk stratification in patients with unstable angina using absolute serial changes of 3 high-sensitive troponin assays. Am Heart J. 2013 Mar;165(3):371-8.e3. doi: 10.1016/j.ahj.2012.11.010. Epub 2013 Jan 24. PMID 23453106
- [Derived] Haaf P, Twerenbold R, Reichlin T, Faoro J, Reiter M, Meune C, Steuer S, Bassetti S, Ziller R, Balmelli C, Campodarve I, Zellweger C, Kilchenmann A, Irfan A, Papassotiriou J, Drexler B, Mueller C. Mid-regional pro-adrenomedullin in the early evaluation of acute chest pain patients. Int J Cardiol. 2013 Sep 30;168(2):1048-55. doi: 10.1016/j.ijcard.2012.10.025. Epub 2012 Nov 27. PMID 23199555
- [Derived] Reichlin T, Twerenbold R, Reiter M, Steuer S, Bassetti S, Balmelli C, Winkler K, Kurz S, Stelzig C, Freese M, Drexler B, Haaf P, Zellweger C, Osswald S, Mueller C. Introduction of high-sensitivity troponin assays: impact on myocardial infarction incidence and prognosis. Am J Med. 2012 Dec;125(12):1205-1213.e1. doi: 10.1016/j.amjmed.2012.07.015. PMID 23164485
- [Derived] Haaf P, Drexler B, Reichlin T, Twerenbold R, Reiter M, Meissner J, Schaub N, Stelzig C, Freese M, Heinzelmann A, Meune C, Balmelli C, Freidank H, Winkler K, Denhaerynck K, Hochholzer W, Osswald S, Mueller C. High-sensitivity cardiac troponin in the distinction of acute myocardial infarction from acute cardiac noncoronary artery disease. Circulation. 2012 Jul 3;126(1):31-40. doi: 10.1161/CIRCULATIONAHA.112.100867. Epub 2012 May 23. PMID 22623715
- [Derived] Potocki M, Reichlin T, Thalmann S, Zellweger C, Twerenbold R, Reiter M, Steuer S, Bassetti S, Drexler B, Stelzig C, Freese M, Winkler K, Haaf P, Balmelli C, Hochholzer W, Osswald S, Mueller C. Diagnostic and prognostic impact of copeptin and high-sensitivity cardiac troponin T in patients with pre-existing coronary artery disease and suspected acute myocardial infarction. Heart. 2012 Apr;98(7):558-65. doi: 10.1136/heartjnl-2011-301269. Epub 2012 Feb 15. PMID 22337952
- [Derived] Schaub N, Reichlin T, Meune C, Twerenbold R, Haaf P, Hochholzer W, Niederhauser N, Bosshard P, Stelzig C, Freese M, Reiter M, Gea J, Buser A, Mebazaa A, Osswald S, Mueller C. Markers of plaque instability in the early diagnosis and risk stratification of acute myocardial infarction. Clin Chem. 2012 Jan;58(1):246-56. doi: 10.1373/clinchem.2011.172940. Epub 2011 Nov 4. PMID 22057876
- [Derived] Reiter M, Twerenbold R, Reichlin T, Benz B, Haaf P, Meissner J, Hochholzer W, Stelzig C, Freese M, Heinisch C, Balmelli C, Drexler B, Freidank H, Winkler K, Campodarve I, Gea J, Mueller C. Early diagnosis of acute myocardial infarction in patients with pre-existing coronary artery disease using more sensitive cardiac troponin assays. Eur Heart J. 2012 Apr;33(8):988-97. doi: 10.1093/eurheartj/ehr376. Epub 2011 Oct 31. PMID 22044927
- [Derived] Hochholzer W, Reichlin T, Twerenbold R, Stelzig C, Hochholzer K, Meissner J, Haaf P, Schaub N, Steuer S, Bassetti S, Reiter M, Roost K, Freidank H, Winkler K, Mueller C. Incremental value of high-sensitivity cardiac troponin T for risk prediction in patients with suspected acute myocardial infarction. Clin Chem. 2011 Sep;57(9):1318-26. doi: 10.1373/clinchem.2011.162073. Epub 2011 Jul 19. PMID 21771945
- [Derived] Reichlin T, Irfan A, Twerenbold R, Reiter M, Hochholzer W, Burkhalter H, Bassetti S, Steuer S, Winkler K, Peter F, Meissner J, Haaf P, Potocki M, Drexler B, Osswald S, Mueller C. Utility of absolute and relative changes in cardiac troponin concentrations in the early diagnosis of acute myocardial infarction. Circulation. 2011 Jul 12;124(2):136-45. doi: 10.1161/CIRCULATIONAHA.111.023937. Epub 2011 Jun 27. PMID 21709058
- [Derived] Reiter M, Twerenbold R, Reichlin T, Haaf P, Peter F, Meissner J, Hochholzer W, Stelzig C, Freese M, Heinisch C, Breidthardt T, Freidank H, Winkler K, Campodarve I, Gea J, Mueller C. Early diagnosis of acute myocardial infarction in the elderly using more sensitive cardiac troponin assays. Eur Heart J. 2011 Jun;32(11):1379-89. doi: 10.1093/eurheartj/ehr033. Epub 2011 Feb 28. PMID 21362702
- [Derived] Hochholzer W, Reichlin T, Stelzig C, Hochholzer K, Meissner J, Breidthardt T, Reiter M, Duehsler B, Freidank H, Winkler K, Twerenbold R, Mueller C. Impact of soluble fms-like tyrosine kinase-1 and placental growth factor serum levels for risk stratification and early diagnosis in patients with suspected acute myocardial infarction. Eur Heart J. 2011 Feb;32(3):326-35. doi: 10.1093/eurheartj/ehq429. Epub 2010 Dec 7. PMID 21138939
- [Derived] Reichlin T, Hochholzer W, Bassetti S, Steuer S, Stelzig C, Hartwiger S, Biedert S, Schaub N, Buerge C, Potocki M, Noveanu M, Breidthardt T, Twerenbold R, Winkler K, Bingisser R, Mueller C. Early diagnosis of myocardial infarction with sensitive cardiac troponin assays. N Engl J Med. 2009 Aug 27;361(9):858-67. doi: 10.1056/NEJMoa0900428. PMID 19710484
- [Derived] Reichlin T, Hochholzer W, Stelzig C, Laule K, Freidank H, Morgenthaler NG, Bergmann A, Potocki M, Noveanu M, Breidthardt T, Christ A, Boldanova T, Merki R, Schaub N, Bingisser R, Christ M, Mueller C. Incremental value of copeptin for rapid rule out of acute myocardial infarction. J Am Coll Cardiol. 2009 Jun 30;54(1):60-8. doi: 10.1016/j.jacc.2009.01.076. PMID 19555842